CLINICAL TRIAL: NCT04585958
Title: A Phase I Study of DS-8201a in Combination With Olaparib in HER2-Expressing Malignancies
Brief Title: Testing the Combination of DS-8201a and Olaparib in HER2-Expressing Cancers With Expansion in Patients With Platinum Resistant Ovarian Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-07841; NCI-2020-07841 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10355 (Other: Dana-Farber - Harvard Cancer Center LAO); 10355 (Other: CTEP); UM1CA186709 (NIH)
Record Dates: First submitted 2020-10-13; First posted 2020-10-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Malignant Solid Neoplasm; Platinum-Resistant Ovarian High Grade Serous Adenocarcinoma; Unresectable Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Biopsy; Specimen Handling; olaparib; trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (trastuzumab deruxtecan, olaparib) (Experimental): Patients receive trastuzumab deruxtecan IV over 30-90 minutes on day 1 and olaparib PO BID on days 1-21, days 8-14, or days 3-9 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. All patients undergo collection of blood samples, ECHO or MUGA, CT, and biopsies throughout the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Drug: Olaparib; Biological: Trastuzumab Deruxtecan

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood and urine samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo echocardiography
  Other Names: EC; Echocardiography
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281
Biological: Trastuzumab Deruxtecan — Given IV
  Other Names: DS-8201; DS-8201a; Enhertu; Fam-trastuzumab Deruxtecan-nxki; T-DXd; WHO 10516

SUMMARY:
This phase I trial identifies the side effects and best dose of DS-8201a and olaparib in treating patients with HER2-expressing cancers that have spread to other places in the body or cannot be removed by surgery or ovarian cancer that remains despite treatment with a platinum treatment (platinum resistant). Olaparib is a drug that blocks an enzyme involved in many cell functions, including the repair of deoxyribonucleic acid (DNA) damage. Blocking this enzyme may help keep tumor cells from repairing their damaged DNA, causing them to die. DS-8201a is an antibody-drug conjugate. This agent has two components: an antibody component and a chemotherapy component. The antibody component is attached to the chemotherapy molecules. Upon administration of DS-8201a, the antibody targets and binds to tumor cells that have abundant HER2 (human-epidermal growth factor receptor 2), which is a protein on the surface of some tumor cells. The chemotherapy then enters the cells and blocks DNA replication in the tumor cells with abundant HER2, causing them to die. Giving DS-8201a and olaparib may shrink or stabilize the cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of the combination of trastuzumab deruxtecan (DS-8201a) in combination with olaparib, and to determine the recommended phase 2 dose (RP2D).

II. To evaluate the safety and tolerability of this combination in a dose expansion cohort in patients with platinum resistant high grade serous ovarian carcinoma.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity as measured by objective response rate (ORR), clinical benefit rate, progression-free survival (PFS), and duration of response (DoR).

II. To measure baseline HER2 expression by immunohistochemistry (IHC) in a central laboratory and correlate with response in the dose escalation and in the dose expansion.

III. To evaluate the plasma pharmacokinetic (PK) profiles of olaparib and DS-8201a metabolites when administered in combination in the dose escalation and in the dose expansion.

IV. To determine markers of DNA damage response (DDR) in tumor specimens at baseline and on-treatment in patients with platinum resistant high grade serous ovarian carcinoma in dose expansion.

EXPLORATORY OBJECTIVES:

I. To measure baseline HER2 expression by immune multiple reaction monitoring-mass spectroscopy (ImmunoMRM), and correlate with baseline central IHC and with response in dose escalation and in dose expansion.

II. To assess the formation of topoisomerase I cleaved complex formation (TOP1cc) in blood specimens and correlate with response in dose escalation and in dose expansion.

III. To assess the formation of TOP1cc in paired on-treatment tumor specimens (after DS-8201a alone and after DS-8201a and olaparib combination) and correlate with response in patients with platinum resistant high grade serous ovarian carcinoma in the expansion.

IV. To measure changes in HER2 expression over the course of treatment by IHC and immune multiple reaction monitoring-mass spectrometry (immunoMRM) and correlate with response in patients with platinum resistant high grade serous ovarian carcinoma in dose expansion.

V. To determine biomarkers of response and resistance in tumor specimens and blood specimens, including whole exome sequencing (WES) and ribonucleic acid (RNA) sequencing.

OUTLINE: This is a dose-escalation study of trastuzumab deruxtecan in combination with olaparib followed by a dose-expansion study.

Patients receive trastuzumab deruxtecan intravenously (IV) over 30-90 minutes on day 1 and olaparib orally (PO) twice daily (BID) on days 1-21, days 8-14, or days 3-9 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. All patients undergo collection of blood samples, echocardiography (ECHO) or multigated acquisition scan (MUGA), computed tomography (CT), and biopsies throughout the trial.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* DOSE ESCALATION PHASE
* Patients must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* Patients must have HER2-positive or HER2-expressing tumors determined by a Clinical Laboratory Improvement Act (CLIA)-certified laboratory. Specific requirement of HER2 status is outlined below:

  * Dose Escalation Module 1 and Module 2:

    * HER2 1-3+ expression by IHC OR
    * HER2 amplification by next generation sequencing panel (NGS) or in situ hybridization (ISH) OR
    * If local testing is not feasible, patients will submit archival tissue for central HER2 testing to determine eligibility. Patients with unknown or negative HER2 testing will not be eligible
  * Dose Escalation Module 3:

    * HER2 1-2+ expression by IHC OR
    * HER2 amplification by next generation sequencing panel (NGS) or in situ hybridization (ISH) OR
    * If local testing is not feasible, patients will submit archival tissue for central HER2 testing to determine eligibility. Patients with unknown or negative HER2 testing will not be eligible
* DOSE EXPANSION PHASE
* Patients must have histologically confirmed platinum resistant, high grade serous ovarian carcinoma. Platinum resistant is defined as radiographic progression < 6 months following the last dose of platinum therapy
* HER2 IHC 1+ per local or central testing
* There must be least one lesion suitable for biopsy without significant risk to the patient
* Patient disease must be evaluable or measurable by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Biopsiable lesion cannot be the only RECIST-measurable lesion
* DOSE ESCALATION AND DOSE EXPANSION PHASES
* Patients must have had at least one prior line of cytotoxic chemotherapy
* Patients can have received an unlimited number of additional lines of chemotherapy, targeted therapy, biologic therapy, or hormonal therapy
* Patients must have archival formalin-fixed paraffin-embedded (FFPE) tissue available for central confirmation of HER2 testing
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of DS-8201a in combination with olaparib in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Hemoglobin >= 10.0 g/dL (within 21 days of randomization/enrollment)

  * No transfusions with red blood cells or platelets are allowed within 1 week prior to screening assessment
* Absolute neutrophil count >= 1,000/mcL (within 21 days of randomization/enrollment)

  * No administration of granulocyte colony-stimulating factor (G-CSF) is allowed within 1 week prior to screening assessment
* Platelets >= 100,000/mcL (within 21 days of randomization/enrollment)

  * No transfusions with red blood cells or platelets are allowed within 1 week prior to screening assessment
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN), (< 3 x ULN in the presence of documented Gilbert's syndrome or liver metastases at baseline) (within 21 days of randomization/enrollment)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN (within 21 days of randomization/enrollment)
* Creatinine =< 1.5 x institutional ULN (within 21 days of randomization/enrollment) OR
* Glomerular filtration rate (GFR) >= 51 mL/min/1.73 m^2 unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73 m^2 (using the Cockcroft-Gault Equation) (within 21 days of randomization/enrollment)
* Patients must have left ventricular ejection fraction (LVEF) >= 50% by either an echocardiogram (ECHO) or multigated acquisition (MUGA) scan within 28 days before randomization/enrollment
* Patients who are human immunodeficiency virus (HIV) positive may participate IF they meet the following eligibility requirements:

  * They must be stable on their anti-retroviral regimen, and they must be healthy from an HIV perspective
  * They must have an undetectable viral load and a CD4 count >= 250 cells/uL within 7 days of enrollment
  * They must not be currently receiving prophylactic therapy for an opportunistic infection and must not have had an opportunistic infection within the past 6 months
  * HIV-infected patients should be monitored every 12 weeks for viral load and CD4 counts
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with brain metastases should be stable and off steroids and at least 4 weeks from radiation at the time of registration
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be better than class 2B
* The effects of DS-8201a and olaparib on the developing human fetus are unknown. For this reason and because HER2 antibody conjugated to a topoisomerase 1 inhibitor agents as well as PARP inhibitors are known to be teratogenic; thus, women of child-bearing potential and men must agree to use highly effective contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for at least 7 months (women of childbearing potential [WOCBP] only) after the last dose of study drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of DS-8201a and olaparib administration
* Women of non-child-bearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases, a blood sample with simultaneous follicle-stimulating hormone [FSH] > 40 mIU/mL and estradiol < 40 pg/mL [< 147 pmol/L] is confirmatory) are eligible. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods outlined for women of child-bearing potential if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method
* Male subjects must not freeze or donate sperm starting at screening and throughout the study period, and at least 4 months after the final study drug administration. Preservation of sperm should be considered prior to enrollment in this study
* Female subjects must not donate, or retrieve for their own use, ova from the time of screening and throughout the study treatment period, and for at least 7 months after the final study drug administration
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible

Exclusion Criteria:

* Patients who have had chemotherapy (including antibody drug therapy) within 4 weeks with the following exceptions: 1 week for weekly paclitaxel; 2 weeks or five half-lives, whichever is longer, for small-molecule targeted agents such as 5-fluorouracil-based agents, folinate agents, hormonal agents; or 6 weeks for nitrosoureas or mitomycin C
* Patients who have had radiation therapy within 4 weeks
* Patients who have had a major surgery within 4 weeks
* Patients who are receiving any other investigational agents
* Patients with a history of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening
* Patients with clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (i.e. pulmonary emboli within three months of the study enrollment, severe asthma, severe chronic obstructive pulmonary disease [COPD], restrictive lung disease, pleural effusion, etc.), and any autoimmune, connective tissue or inflammatory disorders with potential pulmonary involvement (i.e. rheumatoid arthritis, Sjogren's, sarcoidosis, etc.), or prior pneumonectomy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to DS-8201a, the inactive ingredients in the drug product, olaparib, or severe hypersensitivity to other monoclonal antibodies
* Patients receiving any medications or substances that are moderate or strong inhibitors or inducers of CYP3A are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients with a medical history of myocardial infarction within 6 months before randomization/enrollment, symptomatic congestive heart failure (CHF) (New York Heart Association class IIb to IV), troponin levels consistent with myocardial infarction as defined according to the manufacturer 28 days prior to randomization
* Patients with a corrected QT interval (QTc) prolongation to > 470 ms (females) or > 450 ms (males) based on average of the screening triplicate 12-lead electrocardiogram (ECG)
* Patients with multiple primary malignancies within 3 years, except adequately resected non-melanoma skin cancer, curatively treated in-situ disease, and other solid tumors curatively treated
* Patients with an uncontrolled infection requiring IV antibiotics, antivirals, or antifungals
* Patients receiving chloroquine or hydroxychloroquine will require a washout period of >= 14 days to be eligible for the study
* Patients with unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to grade =< 1 or baseline. Subjects with chronic grade 2 toxicities may be eligible per the discretion of the investigator after consultation with the sponsor medical monitor or designee (e.g., grade 2 chemotherapy-induced neuropathy)
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because DS-8201a is a HER2 antibody conjugated to a topoisomerase 1 inhibitor agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with DS-8201a, breastfeeding should be discontinued if the mother is treated with DS-8201a. These potential risks may also apply to other agents used in this study
* Patients who have received a live, attenuated vaccine within 30 days prior to the first dose of DS-8201a

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose/recommended phase 2 dose | Up to 42 days
  Will be measured by Common Terminology Criteria for Adverse Events version (v) 5.0 and analyzed using descriptive statistics.
Incidence of adverse events | Up to 30 days post treatment

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 30 days post treatment
  ORR will be evaluated by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria to determine the best overall response for evaluable patients.
Clinical benefit rate (CBR) | Up to 30 days post treatment
  CBR will be evaluated by RECIST 1.1 criteria to determine the best overall response for evaluable patients.
Duration of response (DOR) | Up to 30 days post treatment
  DOR will be evaluated by RECIST 1.1 criteria to determine the best overall response for evaluable patients. DOR will be described using the method of Kaplan-Meier.
HER2 expression | At baseline
  HER2 expression on archival specimens will be analyzed using current American Society of Clinical Oncology/College of American Pathologists breast cancer and gastric cancer scoring methods. The levels of HER2 expression (0, 1+, 2+, or 3+) will be determined and the number and percentage of patients in each category will be reported. Chi-squared test and regression modeling may be used to investigate any possible relationship of HER2 biomarker levels with anti-tumor efficacy.
Plasma pharmacokinetic (PK) profiles | Up to 30 days post treatment
  PK will be analyzed using descriptive statistics. Analysis of variance and regression model may be used to investigate any possible relationship of PK biomarker levels with anti-tumor efficacy
Markers of deoxyribonucleic acid (DNA) damage response (DDR) | At baseline and on-treatment
  Markers of DDR will be measured by multiplex IF in tumor specimens at baseline and on-treatment in patients with platinum resistant high grade serous ovarian carcinoma in the dose expansion cohort and correlating these markers with response. For the DDR assay, levels exceeding 4% nuclear area positive (NAP) γH2AX, 4% NAP pNBS1, and 5% cells with ≥ 5 Rad51 nuclear foci indicate a DNA damage activation response (Wilsker et al., 2019).

OTHER OUTCOMES:
HER2 expression | Up to 30 days post treatment
  Correlation between HER2 expression, immunohistochemistry (IHC), and response may be evaluated by Chi-squared test and regression model.
Formation of topoisomerase I cleaved complex formation (TOP1cc) in blood samples | Up to 30 days post treatment
  Will measure the formation of formation TOP1cc in blood specimens and correlate with response in the dose escalation and in the dose expansion Will be analyzed using descriptive statistics.
Presence of topoisomerase I cleaved complex formation (TOP1cc) in paired on-treatment tumor specimens | Up to 30 days post treatment
  Will assess the presence of TOP1cc in paired on-treatment tumor specimnes and correlate with response in patients with platinum resistant high grade serous ovarian carcinoma in the dose expansion. Will be analyzed using descriptive statistics.
Changes in HER2 expression | Baseline up to 30 days post treatment
  Will measure changes in HER2 expression over the course of treatment by IHC and immunoMRM and correlate with response in patients with platinum resistant high grade serous ovarian carcinoma in the dose expansion. Will be analyzed using descriptive statistics.
Biomarkers of response and resistance | Up to 30 days post treatment
  Will be analyzed using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth K Lee, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (5):
- United States (5):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm